CLINICAL TRIAL: NCT07048158
Title: Beneficial Effects of "Perfect Heartio" Drink in Improving Cardiovascular Health
Brief Title: "Perfect Heartio" Drink and Cardiovascular Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Perfect Series Sdn Bhd (Industry)
Collaborators: UCSI University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TPH001
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Diseases; Lipid Metabolism Disorders
Keywords: Complementary and alternative medicine; Herbal Medicine
MeSH Terms: conditions — Cardiovascular Diseases; Lipid Metabolism Disorders

STUDY DESIGN:
Intervention Model Description: Subjects will be required to consume Perfect Heartio (PH) drink for 12 weeks, at the dosage of 15g twice daily. Compliance form will be given to monitor the compliance of subject. Assessment will be conducted at week 0, 4, 8 and 12. Perfect Heartio (PH) is a nutritional drink composed of mainly diluted herbal extracts of TCM, including ginger, Glycyrrhiza uralensis, Alternanthera sessilis, Panax notoginseng, Red date, Codonopsis pilosula, Ligusticum chuanxiong, Astragalus membranaceus.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Perfect Heartion Drink Interventional Arm (Experimental): Subjects will be required to consume PH drink for 12 weeks, at the dosage of 15g twice daily. Compliance form will be given to monitor the compliance of subject.
  Interventions: Dietary Supplement: Perfect Heartio Drink

INTERVENTIONS:
Dietary Supplement: Perfect Heartio Drink — Perfect Heartio (PH) drink is a nutritional drink composed of diluted herbal extracts of TCM, including ginger, Glycyrrhiza uralensis, Alternanthera sessilis, Panax notoginseng, Red date, Codonopsis pilosula, Ligusticum chuanxiong, Astragalus membranaceus.

SUMMARY:
Noncommunicable diseases (NCDs) such as type 2 diabetes (T2D) and cardiovascular disease (CVD) account for more deaths globally than any other condition. In 2018, the WHO reported that NCDs accounted for 71% of global deaths. They also showed that low- and middle-income countries are disproportionately affected by NCDs, accounting for 85% of NCD-related deaths among individuals aged 30-69 y. Among NCDs, CVD is the leading and fourth-leading causes of death, accounting for 19.5 million deaths worldwide in 2018. Furthermore, despite increasing global awareness, the prevalence of these conditions continues to increase at alarming rates. Deaths from CVD are expected to reach 23.6 million annually by 2030 from 17.6 million deaths in 2016. The underlying aetiology of these conditions is complex, as they can be influenced by several environmental, genetic, and behavioural factors. However, diet and nutrition play a particularly important role in these conditions, especially in the context of the double burden of malnutrition facing many low- and middle-income countries.

DETAILED DESCRIPTION:
Traditional Chinese Medicine (TCM), one of the intriguing features of traditional Chinese culture, has a history of more than 2,000 years, with both unique theories and rich experience. Because of the lack of objective and quantitative evaluation criteria, TCM is complementary or alternative medicine in most Western countries. However, in China, more than 71.2% of patients who have experienced Western medicine, TCM, and integrative medicine (both Western medicine and TCM) preferred the integrative approach, and 18.7% chose TCM as their favourite. Moreover, TCM is increasingly welcomed in many developed countries, such as Australia and the United States. Importantly, patients who used more types of TCM tended to use much less Western medicine recommended by current guidelines. Recent review also highlighted the potential use of TCM as a complementary and alternative approach to the primary and secondary prevention of cardiovascular disease. Perfect Heartio (PH) is a nutritional drink composed of mainly diluted herbal extracts of TCM, including ginger, Glycyrrhiza uralensis, Alternanthera sessilis, Panax notoginseng, red date, Codonopsis pilosula, Ligusticum chuanxiong, Astragalus membranaceus. Broad pharmacological properties of ginger and its bioactive components have been reported, suggesting its potential use in preventing CVD. Glycyrrhiza uralensis stands out for its exceptional therapeutic potential, particularly in enhancing cardiac muscle regeneration, and slowing muscle aging. Alternanthera sessilis has been showed to prevent cardiovascular and liver diseases. Panax notoginseng improve angiogenesis. Red date exerts anti-adipogenicity effects and enhancing endothelial function. Codonopsis pilosula improves the functional state of the cardiovascular system and mitigating the onset and progression of CVD. Ligusticum chuanxiong has been showed to promote blood circulation and remove blood stasis. Astragalus membranaceus also showed to improve cardiovascular function, protect myocardial cells, and increase coronary blood flow.

ELIGIBILITY:
Inclusion Criteria:

* General healthy subjects during enrolment
* Age 18 and above
* Willing to comply with interventional plan and comes to do follow up
* Willing to gives consent

Exclusion Criteria:

* Use nonsteroidal anti-inflammatory drugs (NSAIDs) more than once a week during enrolment
* Use of anticoagulants or corticosteroids
* Use of individual supplements of vitamin A, E, or beta carotene more than once a week during enrolment
* Renal failure or dialysis, cirrhosis, other serious conditions that precluded participation
* No previous history of cancer (except nonmelanoma skin cancer)
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Lipid profile | Week 0, 4, 8 and 12
  Total cholesterol levels, Triglycerides levels, LDL- cholesterol levels, HDL-cholesterol levels
Cardiac inflammatory levels | Week 0, 4, 8 and 12
  C-reactive protein
Cardiac injury levels | Week 0, 4, 8 and 12
  Creatine kinase
Cardiac remodelling status | Week 0, 4, 8 and 12
  Matrix metalloproteinases-9 (MMP-9)

SECONDARY OUTCOMES:
Quality of Life of subject | Week 0, 4, 8 and 12
  Scale title: HeartQoL (Heart-related Quality of Life questionnaire). Minimum and maximum values: ranges from 0 to 3. Interpretation: Higher scores indicate better health-related quality of life. The global score is the mean of all answered items (14 total: 10 physical and 4 emotional).
Self-perceived health status | Week 0, 4, 8 and 12
  Scale title: Visual Analogue Scale (VAS). Minimum and maximum values: 0 to 10. Interpretation: Higher scores indicate better cardiovascular health. In this context, a score of 0 represents the worst imaginable cardiovascular health, while a score of 10 represents the best imaginable cardiovascular health as perceived by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Chung Keat Tan, PhD, Principal Investigator — UCSI University
Locations (1):
- UCSI University, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study are available from the corresponding author on reasonable request. All of the individual participant data collected during the trial, after de-identification will be shared upon reasonable request. Additional documents including study protocol, statistical analysis plan, informed consent form and clinical study report will also be made available. The data will be available immediately following publication with no end date. Data will be shared with anyone who wishes to access with reasonable request. The data can be used for any types of analyses.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon publication of the study outcomes, for a time frame of 5 years
Access Criteria: The datasets generated during and/or analysed during the current study are available from the corresponding author on reasonable request. All of the individual participant data collected during the trial, after de-identification will be shared upon reasonable request. Additional documents including study protocol, statistical analysis plan, informed consent form and clinical study report will also be made available. The data will be available immediately following publication with no end date. Data will be shared with anyone who wishes to access with reasonable request. The data can be used for any types of analyses.

REFERENCES:
- [Background] Cooper F. How to publish a winning newsletter. Health Care Can. 1979 Sep;21(9):41-2. No abstract available. PMID 10243891
- [Background] Ling Lee W, Chinna K, Sumintono B. Psychometrics assessment of HeartQoL questionnaire: A Rasch analysis. Eur J Prev Cardiol. 2021 Oct 13;28(12):e1-e5. doi: 10.1177/2047487320902322. Epub 2020 Feb 4. No abstract available. PMID 34647582